CLINICAL TRIAL: NCT05028920
Title: The Study on Nutritional Status of Patients With Mild Cognitive Impairment
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 201900610B0
Record Dates: First submitted 2021-06-23; First posted 2021-08-31 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The global aging population is rising year by year. According to the result of Taiwan epidemiological survey, dementia has become the health issue in aging population. Mild cognitive function impairment may present years before dementia is diagnosed. Therefore early diagnosis of dementia at its Mild cognitive function impairment stage is beneficial for disease prevention and potentially delaying the deterioration of cognitive function impairment. Nutritional status includes a healthy diet, favor body composition and activity habits, which not only reduces the risk of nutritional metabolic diseases, but also has a direct relationship with delaying cognitive function impairment. The dietary quality index of Mediterranean-Dietary Approaches to Stop Hypertension Intervention for Neurodegenerative Delay diet (MIND diet) may prevent aging and positively associated with delaying dementia in elderly. However, the result in dietary quality index and delaying cognitive function impairment from current studies were still unclear. In additions, based on the differences in dietary patterns between Taiwan and Western countries, no current calorie and dietary nutrition recommendations. This cross-sectional study is to investigate the association between dietary quality index and nutritional status risk factors in cognitive function impairment patients and expected to develop an assessment tool for Taiwanese clinical nutrition strategies and applications.

DETAILED DESCRIPTION:
Aging populations is rising by years in Taiwan. Mild cognitive function impairment (MCI) has become the important health issue. Current knowledge of the etiology of cognitive decline is incomplete, the potential modifiable factors, such as diet may delay the deterioration of disease. This study is aimed to comprise the differences nutritional status,include dietary nutrients intake, MIND diet scores,body composition analysisin with mild cognitive impairment. Design and methods: this cross-sectional study from July, 2019. According to clinical dementia rating (CDR) and mini-mental state examination (MMSE), subjects are divided into healthy group (CDR = 0 and MMSE ≧ 26) and MCI group (CDR ≧ 0.5 and MMSE ≧ 26). Dietary data were obtained by 3-day dietary records and nutrients intake were calculated by trained dietitian. We expected to understand the nutritional status of patients with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥40 years old (regardless of gender)
2. Complete 3-day dietary record, Mini-mental state examination and Clinical dementia rating assessment
3. Independent physical activity

Exclusion Criteria:

1. No amputation, edema, cancer, terminal case, thyroid disease and stroke include stroke history
2. No family support
3. Psychological problem
4. Extremely data of dietary record(< 500 kcal or > 3500 kcal)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild cognitive function impairment (MCI) may present years before dementia is diagnosed. Therefore early diagnosis of dementia at its MCI stage is beneficial for disease prevention and potentially delaying the deterioration of cognitive function impairment.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The dietary quality index: Mediterranean-DASH Intervention for Neurodegenerative Delay diet | at the 12th month
  The MIND score is based on 10 brain-healthy foods groups: namely, higher intake of green leafy vegetables (spinach, lettuce, kale), other vegetables,berries(blueberries,strawberries), nuts, whole grains, fish, beans, poultry, limited intake of wine (red and white wine), and use of olive oil as primary source of fat; and 5 unhealthy foods: namely, lower intakes of butter and margarine, cheese, red meat and products, fast fried foods, and pastries and sweets.For healthy components, assigned 0, 0.5 or 1 point for higher intakes, and for unhealthy components the scoring was reversed (total score 0 to 15 points).
Assessment cognitive function only one time: Mini-mental state examination scale, MMSE | at the 1st month
  Assessment tools of cognitive impairment.Scores: 0 - 30 points. Among the result of MMSE=23.5±6.6(p<0.05)
Assessment cognitive function only one time:Clinical dementia rating scale, CDR | at the 1st month
  Assessment tools of cognitive impairment.Scores: 0 - 5 points(0 points for normal,0.5 points for mild cognitive impairment, 1 points for mild dementia, 2 points for moderate dementia, 3 points for severe dementia).
  Among the result of CDR=0.4±0.5(p<0.05)

SECONDARY OUTCOMES:
Lipid profile | at the 1st,12th month
  Serum HDL-Cho, LDL-Cho, triglyceride and total cholesterol are in milligram per deciliter
Kidney function | at the 1st,12th month
  Serum BUN,Creatine and urine acid are in milligram per deciliter
Liver function | at the 1st,12th month
  Serum AST,ALT and bilirubin-total are in units per liter.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan